CLINICAL TRIAL: NCT04855487
Title: Assessing the Feasibility, Acceptability, and Preliminary Efficacy of an Expressive Storytelling Intervention for Adolescents and Young Adults With Cancer to Share Stories With Oncology Nurses
Brief Title: Expressive Storytelling to Share Adolescents/Young Adults Cancer Stories
Acronym: ESSAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Eunji Cho, Postdoctrol Fellow, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VR55572
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Pediatric Cancer; Growth, Posttraumatic; Nurse-Patient Relations; Narrative Medicine
Keywords: Storytelling; Adolescents and young adults with cancer; Nursing intervention; Human flourishing; Resilience
MeSH Terms: conditions — Neoplasms; Narrative Medicine

STUDY DESIGN:
Intervention Model Description: Adolescents/young adults with cancer will participate in a 5-week online expressive storytelling intervention. They will independently create digital stories about themselves while their target audiences are their primary nurses. They will then participate in weekly online meetings with nursing research staff, during which they introduce their stories and discuss their reflections. In the final session, they will create a one-page or five-slide story to share with their primary nurses, if they want.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Adolescents/young adults with cancer will participate in a 5-week online expressive storytelling intervention. They will independently create digital stories about themselves while their target audiences are their primary nurses. They will then participate in weekly online meetings with nursing research staff, during which they introduce their stories and discuss their reflections. In the final session, they will create a one-page or five-slide story to share with their primary nurses, if they want.
  Interventions: Behavioral: Nurse-patient dyadic storytelling intervention

INTERVENTIONS:
Behavioral: Nurse-patient dyadic storytelling intervention — During the 5-week online intervention, adolescents/young adults with cancer will create their stories following the guiding questions and online meetings with nursing research staff. The target audience of their stories will be their primary nurses. This online dyadic storytelling intervention is designed to promote in-depth self-reflection and meaningful and therapeutic relationships within bedside nurses. The intervention is designed following the Story Theory and Pennebaker's Expressive Writing paradigm.

SUMMARY:
The purpose of this study is to test the feasibility, acceptability, and preliminary efficacy of an online expressive storytelling intervention for adolescents and young adults (AYA) with cancer.

* Specific Aim 1. To evaluate the feasibility and acceptability of a 5-week online expressive storytelling intervention. We will (a) conduct a 1-group pre- and post-test study with 20 AYA with cancer and (b) examine feasibility and acceptability through study enrollment rates, retention rates, usability score, adherence and data collection rates, satisfaction score, perceived benefits score, and intervention fidelity.

  *Hypothesis 1: We will reach following feasibility and acceptability benchmarks: (a) >70% enrollment of eligible participants, (b) >70% retention, (c) >75% adherence and data collection, (d) >70 out of 100 usability score, (e) >5 out of 7 satisfaction score, (f) >average 5 on the perceived benefits score, and (g) >3 out of 4 fidelity score.
* Specific Aim 2. To assess preliminary efficacy of a 5-week online expressive storytelling intervention.

  * Hypothesis 2: AYA participants will report lower psychosocial distress, higher health-related quality of life, and higher well-being scores postintervention.

DETAILED DESCRIPTION:
* Rationale/Significance of Study: Cancer is one of life's most stressful and serious illnesses for adolescents and young adults (AYA). In 2021, approximately 15,000 AYA ages 15 to 25 years are expected to be newly diagnosed with cancer in the United States. Despite high survival rates exceeding 85%, the burden of cancer and its' treatment for AYA is substantial and prolonged due to their unique developmental characteristics. AYA with cancer often deal with the difficulties of transition from pre-cancer to treatment trajectory while also transitioning from adolescence to young adulthood. While they suffer from physical, emotional, psychosocial, and financial burdens as a result of cancer, establishing resources for future development and well-being, such as identity and goal development, education, and social relationships, often becomes secondary during treatment because of concerns about survival. As a result, AYA with cancer have less opportunities to be prepared for their lifelong challenges and build abilities to deal with such complex suffering, which lead to maladjustment, hinder social reintegration, and limit their ongoing well-being. Thus, there is a critical need to deliver developmentally appropriate supportive care for AYA with cancer to reduce the potential risk of negative consequences and improve capacities to thrive throughout their life trajectories. The proposed study aims to test the feasibility, acceptability, and preliminary efficacy of an expressive storytelling intervention for AYA with cancer, helping them create and share their stories.
* Theoretical Framework: The theoretical framework of our study and the intervention contents are designed following the Story Theory in nursing practice and the Self-transcendence Theory. Our intervention development process follows the Obesity-Related Behavioral Intervention Trials (ORBIT) model to develop and evaluate complex interventions.
* Design and Procedures: A single-group pre- and post-test clinical trial design will be applied. A total of 20 dyads of AYA with cancer will be recruited. Each AYA will be asked to think of three to five of their primary nurses as audiences of their stories created during the 5-week online storytelling intervention. The AYA participant will create digital stories about themselves following the guiding questions. The dyad will then participate in weekly online meetings with nursing research staff, during which they will introduce their stories and discuss their reflections. Participants will complete pre- (T1) and post-intervention (T2) measures and share their qualitative feedback.
* Implications for Practice: Results will serve as the foundational knowledge to conduct a large-scale, randomized clinical trial. Ultimately, this study will promote well-being and improve palliative and psychosocial nursing care to individuals with serious illness, including AYA with cancer.

ELIGIBILITY:
[Inclusion Criteria] 1.1 AYA ages 15 to 25 years. Age criterion was determined based on (a) the age criteria of adolescence (15-17 years) and emerging adulthood (18-25 years) guided by lifespan developmental frameworks35 and (b) the intervention being developmentally appropriate for this unique age group.

1.2 Patients must have any type of histologically or cytologically confirmed malignancy during adolescence or young adulthood.

1.3 Patients may be at any stage of the cancer trajectory. Participants can be enrolled beginning one month after an initial cancer diagnosis.

1.4 Patients must be cognitively intact.

1.5 Patients must have access to the internet using their own electronic devices (e.g., laptop, desktop, tablet PC, smartphone).

1.6 Ability to speak, write, read, understand English.

[Exclusion Criteria] 2.1 Patients who have any unanticipated needs that cannot be accommodate by the PI (e.g., technical challenges, permanent loss of electronic devices, permanently unable to access the internet) can be excluded before and during the participation.

2.2 Patients who show their unwillingness to participate in the program by their actions (e.g., providing false information, just giggling rather than answering questions, increases in aggression or anxiety) can be discussed to make a decision about honoring their desire to withdraw from participation.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Secure Flourish Measure (Adolescent Version) | Day 0, Day 35
  A 12-item 10-point Likert scale measure ranging from 0 (Not Satisfied at Aall) to 10 (Completely Satisfied) to assess adolescents' level of human flourishing. This measure is tailored to adolescents (12-18 years old).
Change in Secure Flourish Measure (Adult Version) | Day 0, Day 35
  A 12-item 10-point Likert scale measure ranging from 0 (Not Satisfied at All) to 10 (Completely Satisfied) to assess young adults' level of human flourishing. This measure is tailored to individuals over 18 years old.
Change in Herth Hope Index Scale | Day 0, Day 35
  A 12-item 4-point Likert scale measure ranging from 1 (Strongly Disagree) to 4 (Strongly Agree) to assess hope in adolesents and young adults with cancer.
Change in Perceived Social Support from Health Care Professionals | Day 0, Day 35
  A 20-item 5-point Likert scale measure ranging from 1 (Totally Disagree) to 5 (Totally Agree) to asess adolescent/young adults' perceived social support from health care providers
Change in Self-transcendence Scale | Day 0, Day 35
  A 15-item 4-point Likert scale measure ranging from 1 (Not at All) to 4 (Very Much) to assess the level of self-transcendence in adolescents/young adults with cancer
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v. 2.1 (Adult Version) | Day 0, Day 35
  A measure consists of 28 5-point Likert scale items and one 11-point Likert scale item (asking about general pain) to assess the self-perceived health related quality of life in young adults with cancer
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) 25 v. 2.0 (Adolescent Version) | Day 0, Day 35
  A measure consists of 24 5-point Likert scale items and one 11-point Likert scale item (asking about general pain) to assess the self-perceived health related quality of life in adolescents with cancer
Satisfaction Survey | Day 35
  A 16-item survey to assess participants' satisfaction of the intervention program. Ten 7-point Likert scale items assess satisfaction, and 6 items assess perceived benefits of the intervention.
System Usability Survey | Day 35
  A 10-item survey to assess participants' perceived usability of the intervention program. This scale uses 5-point Likert scale (range from Strongly Agree to Strongly Disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Eunji Cho, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
There are no tangible resources to share at this time as the intervention is in testing phases. We plan to make the intervention available for sharing in the future, upon completed testing. Therefore, data is the only resource available for sharing.
  The proposed research will produce data with 20 adolescent/young adult with cancer. The final data set will contain (a) demographic information, (b) feasibility and acceptability information, and (c) preliminary efficacy of the online expressive storytelling intervention on the well-being in adolescents and young adults with cancer.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available for sharing no later than the publication date of the main results from the final dataset. Data will be disclosed without a specific deadline.
Access Criteria: The data will be shared with anyone who is interested in this study. We especially seek to make our data available to the community of scientists interested in adolescent and young adult oncology and psychosocial interventions utilizing the power of narratives and nurse-patient therapeutic relationships.